CLINICAL TRIAL: NCT03086993
Title: Randomized, Controlled Study to Compare the Efficacy, Safety and Pharmacokinetics of Melphalan/HDS Treatment Given Sequentially Following Cisplatin/Gemcitabine Versus Cisplatin/Gemcitabine in Patients With IntraHepatic Cholangiocarcinoma
Brief Title: Percutaneous Hepatic Perfusion vs. Cisplatin/Gemcitabine in Patients With Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHP-ICC-203
Record Dates: First submitted 2017-03-13; First posted 2017-03-22 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Bile Duct Cancer; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Cholangiocarcinoma | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melphalan/PHP (Experimental): Patients may receive up to 6 treatments of Melphalan/HDS 3.0 mg/kg IBW. Each treatment cycle consists of 6 weeks with an acceptable delay for an additional 2 weeks (i.e. 8 weeks in total). The maximum dose of melphalan will be 220 mg per treatment.
  Interventions: Combination Product: Melphalan/HDS
- Cisplatin and Gemcitabine (Active Comparator): Each Cis/Gem treatment cycle will comprise cisplatin, dosed at 25 mg per square meter of body surface area, and gemcitabine, dosed at 1000 mg per square meter of body surface area. Each will be administered on Days 1 and 8 every 3 weeks.
  Interventions: Drug: Cisplatin and Gemcitabine

INTERVENTIONS:
Combination Product: Melphalan/HDS — Melphalan/HDS treatment for up to six cycles, followed by a re-induction of CisGem.
  Other Names: Melphalan/PHP
  Arms: Melphalan/PHP
Drug: Cisplatin and Gemcitabine — continuous treatment with Cis/Gem until disease progression
  Other Names: Cis/Gem
  Arms: Cisplatin and Gemcitabine

SUMMARY:
This study will evaluate two groups of patients who have intrahepatic cholangiocarcinoma. Each group will receive induction treatment with Cisplatin and Gemcitabine per SOC for 4 treatment cycles. Following induction treatment patients will be randomize (1:1), to 2 arms of treatment. One group (50%) will be receive high dose chemotherapy delivered specifically to the liver, while the other group (50%) will continue treatment with Cisplatin and Gemcitabine. Patient in each group will get repeating cycles of treatment until the cancer advances. All patients will be followed until death. This study will compare the overall survival (OS) in patients with intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
The study will consist of 4 phases: a screening, an induction, randomization and follow-up phase.

Screening phase: Screening assessments will be conducted within 28 days prior to initiation of Induction Phase treatment to determine each patient's overall eligibility. These assessments will include medical history; physical examination; Eastern Cooperative Oncology Group (ECOG) performance status (PS); 12 lead electrocardiogram (ECG); echocardiogram (ECHO); vital signs; laboratory assessments; radiologic assessments of disease status; and an evaluation of the vasculature compatibility for Percutaneous Hepatic Perfusion (PHP).

Induction phase: The initial 12 weeks of the study, all patients will receive 4 cycles of cisplatin/gemcitabine. Each cycle will be comprised of cisplatin dosed at 25 mg per square meter of body-surface area (BSA), followed by gemcitabine dosed at 1000 mg per square meter of BSA; dosing will occur on Days 1 and 8 of each cycle. At the completion of 3 cycles (week 8 (+1 week)) of cisplatin/gemcitabine, an imaging scan is performed as per standard of care to determine if the patient has progressed on treatment or should continue receiving the cisplatin/gemcitabine induction therapy for one more cycle (4th cycle - prior to randomization). At the completion of 4 cycles (week 12 (+1 week)) of cisplatin/gemcitabine, patients will undergo whole-body imaging to determine the status of their disease. Patients with progressive disease (PD) will be discontinued from study treatment, and will receive further treatment to be determined by the principal investigator (PI). They will continue to be followed until death or the end of the study. Patients who have at least stable disease (SD) at imaging after induction phase of 4 cycles of cisplatin/gemcitabine (week 12 (+ 1 week)) will go on to the next phase of the study (Randomized Treatment Phase).

Randomization phase: Patients who have at least stable disease via imaging at the end of the Induction Phase will be randomized in a 1:1 ratio to Melphalan/HDS treatment or to continue cisplatin/gemcitabine in cycles previously described in the Induction Phase, until progressive disease (PD) or unacceptable toxicity is observed. Patients who were randomized to treatment with Melphalan/HDS (dosed at 3.0 mg/kg Ideal Body Weight [IBW]) must undergo their first treatment within 14 days following the whole body imaging performed at end of the Induction Phase. For Melphalan/HDS treatment, patients will receive up to 6 treatments. Each treatment cycle will consist of 6 weeks with an acceptable delay for up to another 2 weeks before the next planned treatment to allow for additional recovery, if needed. After the Melphalan/HDS treatment, in the absence of disease progression, the patient should undergo a re-induction of CisGem. Tumor response will be assessed in both treatment arms every 8 weeks (+ 1 week) until PD.

The assessment scans will be reviewed by Independent Review Committee (IRC). At any time when PD is observed, the patient will be removed from further study treatment; any further treatment will be at the discretion of the investigator. Melphalan/HDS treatment will also be discontinued in the event that recovery requires more than 8 weeks from last treatment. An end-of-treatment visit will be conducted approximately 6 to 8 weeks following the final dose of study treatment. Ongoing adverse events (AEs) at the end-of-treatment visit will be followed until the severity returns to common terminology criteria for adverse events (CTCAE) Grade < 1.

Follow-up phase: In the event that disease has not progressed at the end-of-treatment visit, disease assessment scans will continue every 8 weeks (+ 1 week) until PD is documented. Patients will be contacted by phone every 6 months for survival status for the first two years following the completion of study treatment, then yearly thereafter until death, withdrawal of informed consent or they become lost to follow-up, whichever occurs first. Patients will be monitored for two years following the completion of study treatment for the development of myelodysplasia and secondary leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to provide signed informed consent.
2. Intrahepatic cholangiocarcinoma diagnosed by histology.
3. Unresectable ICC, with less than 50% of the liver involved, and without clinically significant extra-hepatic disease (regional lymph node lesions [≤ 2 cm] are acceptable) based on CT
4. Scans used to determine eligibility (CT scan of the chest/abdomen/pelvis and liver) must be performed within 28 days prior to initiation of Induction Phase treatment.
5. At least one target lesion based on the evaluation criteria in solid tumors (RECIST 1.1).
6. Patients must have an ECOG PS of 0-1 at screening.
7. Male or female patients aged ≥ 18 years.
8. Patients must weigh ≥ 35 kg (due to possible size limitations with respect to percutaneous catheterization of the femoral artery and vein using the Delcath Hepatic Delivery System).

Exclusion Criteria:

1. Greater than 50% tumor burden in the liver by imaging.
2. History of orthotopic liver transplantation, hepatic vasculature incompatible with perfusion, hepatofugal flow in the portal vein or known unresolved venous shunting. Prior Whipple procedure is permitted provided the anatomy is still compatible for perfusion with the Melphalan/HDS system.
3. History of, or known, hypersensitivity to any components of melphalan or the components of the Melphalan/HDS system.
4. History of, or known, hypersensitivity to gemcitabine or platinum-containing compounds.
5. Known hypersensitivity to heparin or the presence of heparin-induced thrombocytopenia.
6. Prior treatment with gemcitabine or platinum-containing compounds, including in the adjuvant setting.
7. Received an investigational agent for any indication within 30 days prior to first treatment.
8. Prior radiation therapy to the liver including 90Y , I131 based loco regional therapy. Prior loco regional therapy, including resection, based on other technology for ICC, if any, must have been completed at least 4 weeks prior to baseline imaging.
9. Not recovered from side effects of prior therapy to ≤ Grade 1 (according to National Cancer Institute [NCI] CTCAE version 4.03). Certain side effects that are unlikely to develop into serious or life-threatening events (e.g. alopecia) are allowed at > Grade 1.
10. Those with New York Heart Association functional classification II, III or IV; active cardiac conditions including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), worsening or new-onset congestive heart failure, significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia.
11. History or evidence of clinically significant pulmonary disease that precludes the use of general anesthesia.
12. Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator, makes it undesirable for the patient to participate in the trial (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease).
13. Patients with active bacterial infections with systemic manifestations (malaise, fever, leukocytosis) are not eligible until completion of appropriate therapy. Patients taking low-dose antibiotics for biliary obstruction are exempted from this exclusion criterion.
14. History of prior malignancy that will interfere with the response evaluation (exceptions include in-situ carcinoma of the cervix treated by cone-biopsy/resection, non-metastatic basal and/or squamous cell carcinomas of the skin, any early stage (stage I) malignancy adequately resected for cure greater than 5 years previously).
15. Acute or active hepatitis B or hepatitis C infection. Patients with anti-hepatitis B core antigen (HBc) positive, or hepatitis B surface antigen (HBsAg) but viral deoxyribonucleic acid (DNA) negative are exception(s).
16. History of bleeding disorders which would put a patient at risk for bleeding with anti-coagulation or patients with an increased risk of thromboembolic or hemorrhagic events (e.g., stroke).
17. Brain lesions or intracranial abnormalities at risk for bleeding, by history or radiologic imaging (e.g., active metastases).
18. Known varices at risk of bleeding, including medium or large esophageal or gastric varices, or active peptic ulcer.
19. Inadequate hematologic function as evidenced by any of the following:

    1. Platelets < 100,000/µL
    2. Hemoglobin < 10.0 g/dL, independent of transfusion or growth factor support
    3. White blood cell count (WBC) < 2,000/µL
    4. Neutrophils < 1,500 cells/µL.
20. Serum creatinine > 1.5 mg/dL. If serum creatinine > 1.5 mg/dL, the measured creatinine clearance must be measured and patient is eligible if creatinine clearance > 45 mL/min.
21. Inadequate liver function as evidenced by any of the following:

    1. Total serum bilirubin > 1.5 times ULN
    2. Aspartate aminotransferase (AST) > 5 times the upper limit of normal (ULN) or alanine aminotransferase (ALT) > 5 times ULN
    3. Serum albumin < 2.9 g/dL.
22. Known alcohol or drug abuse that would preclude compliance with study procedures.
23. For female patients of childbearing potential (defined as having had a menstrual period within the past 12 months): a positive serum pregnancy test (β-human chorionic gonadotropin [β HCG]) within 7 days prior to enrollment; or unwilling or unable to undergo hormonal suppression to avoid menstruation during treatment; or if breastfeeding, unwilling or unable to stop breastfeeding while on study treatment.
24. Sexually active females of childbearing potential and sexually active males with partners of reproductive potential: unwilling or unable to use appropriate contraception from screening until at least 6 months after last administration of study treatment.
25. Patients taking immunosuppressive drugs or who are unable to be temporarily removed from chronic anti-coagulation therapy.
26. Patients with biliary stents.
27. Patients with a history of external percutaneous transhepatic cholangiography catheter placement.
28. Patients previously treated with any intra-arterial regional hepatic therapy such as trans-arterial chemoembolization.
29. Patients with severe allergic reactions to iodine contrast which cannot be controlled by premedication with antihistamines and steroids.
30. Patients with a latex allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Change in survival is being assessed through study completion, an average of 2 years
  Patients will be followed until death

SECONDARY OUTCOMES:
Progression-free survival, as determined by IRC | Change in PFS change will be assessed every 9 weeks through study completion, an average of 1 year
  Period of time from 1st treatment to tumor progression or death
Objective response rate (CR + PR) as determined by the Investigator | ORR change will be assessed every 9 weeks through study completion, an average of 1 year
  The number of patients with either a complete or partial response as determined by the investigator

OTHER OUTCOMES:
Progression-free survival, as determined by the Investigator | PFS change will be assessed every 9 weeks through study completion, an average of 1 year
  Period of time from 1st treatment to tumor progression
Objective response rate as determined by IRC | ORR change will assessed every 9 weeks through study completion, an average of one year
  The number of patients with either a complete or partial response as determined by the IRC
Quality of Life (QOL) as measured by the functional health survey EQ-5D module | QOL change will be evaluated every 6 weeks through study completion, an average of 1 year
  QoL will be evaluated for all patients treated in the study
Pharmacokinetic Outcome Measures: Cmax | PK is assessed at each Melphalan/HDS cycle approximately every 6 weeks for an average of one year
  Observed maximum concentration (Cmax)
Pharmacokinetic Outcome Measures: AUC | PK is assessed at each Melphalan/HDS cycle approximately every 6 weeks for an average of one year
  Area under the curve (AUC)
Pharmacokinetic Outcome Measures: Tmax | PK is assessed at each Melphalan/HDS cycle approximately every 6 weeks for an average of one year
  Time of maximum concentration (Tmax)
Pharmacokinetic Outcome Measures: CL | PK is assessed at each Melphalan/HDS cycle approximately every 6 weeks for an average of one year
  Total system clearance (CL)
Incidence of Treatment-Emergent Adverse Events (Safety) | Adverse events are assessed from time of informed consent through the study completion, average about 1 year
  Number of patients experiencing treatment related adverse events as assessed by CTCAE version 4.0

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Duke Health, Durham, North Carolina
  - Ohio State University/Teaching Hospital, Columbus, Ohio
  - West Cancer Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No